CLINICAL TRIAL: NCT05642000
Title: The Safer At School Early Alert HUB
Acronym: SASEA HUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rebecca Fielding-Miller, Assistant Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1U01HD108787-01 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SASEA HUB (Experimental): Access to online COVID-19 information tool hub to support testing access
  Interventions: Behavioral: SASEA HUB
- Control (No Intervention)

INTERVENTIONS:
Behavioral: SASEA HUB — SASEA HUB website, an intervention tool to increase COVID-19 testing
  Arms: SASEA HUB

SUMMARY:
Schools serve important community roles beyond academic education. In historically marginalized communities they are trusted providers for a range of support services for families in need. The tradeoff between these crucial benefits of in-person learning against the risk of SARS-CoV-2 transmission in school settings has been hotly debated throughout much of 2020 and 2021. The stakes are particularly high in historically marginalized communities which rely most heavily on school services, but have also been hit the hardest by COVID-19 primarily due to structural issues. The Safer at School Early Alert (SASEA) program was co-developed by the University of California, San Diego, the County of San Diego, and 15 partner schools serving socially vulnerable students in 5 school districts across San Diego County. SASEA utilizes daily wastewater and surface (floor) environmental monitoring to detect asymptomatic SARS-CoV-2 infections among students and staff on campus. Positive environmental signals are immediately followed by targeted responsive testing for a whole school (in the case of wastewater) or classroom (for a positive surface sample). In this project, we will develop the Safer at School Early Alert HUB (SASEA HUB), an online school environmental monitoring report dashboard with resources to address structural barriers to COVID-19 diagnostic testing in historically marginalized communities (Aim 1). We will also create a toolkit to allow any school to rapidly adapt the template to their specific setting. In Aims 2 and 3, we will use a randomized stepped wedge trial to compare SASEA (control) vs SASEA HUB (intervention) in 26 schools across 3 diverse school clusters in San Diego County. Our primary outcome (Aim 2) is higher rates of diagnostic testing in intervention schools. Our secondary outcome (Aim 3) is increased risk mitigation behaviors in school community members when environmental surveillance data suggests a potential case on campus. In Aim 4, we will use parent-child narrative interviews with 40 parent-student pairs to understand how children perceive COVID-19 risk at school, assess differences in perceptions of testing barriers between intervention and control sites, and better understand how children understand the process of environmental surveillance and responsive testing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 18 and above affiliated with students attending the 3 school districts participating in the SASEA study

Exclusion Criteria:

* Children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only parents were considered enrolled in the study. Staff who were also parents of children who attended the school were also recruited to complete the survey but they are completing the survey in their role as a parent and not as a staff of the school
Units Other Than Participants: schools
Groups:
- Cluster 1: SASEA HUB intervention after 2 week baseline data collection. 12 weeks of intervention exposure.
- Cluster 2: SASEA HUB intervention arm after 2 weeks of baseline data collection (district began fall term two weeks later than Cluster 1). 10 weeks of intervention exposure
- Cluster 3: SASEA HUB intervention after 6 weeks of baseline data collection. 8 weeks of intervention exposure
Period: Wave 1: Late September
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 67; 11 schools | 38; 7 schools (School started a week late for this cluster therefore they did not participate in the first wave of surveys) | 39; 8 schools
Completed | 67; 11 schools | 38; 7 schools | 39; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools
Period: Wave 2: Early October
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 52; 11 schools | 50; 7 schools | 42; 8 schools
Completed | 52; 11 schools | 50; 7 schools | 42; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools
Period: Wave 3: Late October
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 85; 11 schools | 54; 7 schools | 55; 8 schools
Completed | 85; 11 schools | 54; 7 schools | 55; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools
Period: Wave 4: Early November
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 51; 11 schools | 24; 7 schools | 54; 8 schools
Completed | 51; 11 schools | 24; 7 schools | 54; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools
Period: Wave 5: Mid November
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 71; 11 schools | 24; 7 schools | 54; 8 schools
Completed | 71; 11 schools | 24; 7 schools | 54; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools
Period: Wave 6: Early December
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 70; 11 schools | 93; 7 schools | 33; 8 schools
Completed | 70; 11 schools | 93; 7 schools | 33; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools
Period: Wave 7: Late December
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3
Started | 17; 11 schools | 35; 7 schools | 21; 8 schools
Completed | 17; 11 schools | 35; 7 schools | 21; 8 schools
Not Completed | 0; 0 schools | 0; 0 schools | 0; 0 schools

BASELINE CHARACTERISTICS:
Population: This was a stepped-wedge trial. Participants all started as controls and crossed over to the intervention - SASEA HUB
Groups:
- Control: School specific standard of care for COVID-19
- Total: Total of all reporting groups
Arm/Group | SASEA HUB | Control | Total
Number analyzed (Participants) | 917 | 0 | 917
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (6.7) |  | 35.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 809 |  | 809
  Male | 108 |  | 108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 917 |  | 917

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Completed a COVID-19 Test
Description: The primary study endpoint will be student diagnostic testing uptake in the previous 14-days, measured using household surveys distributed at 2-week intervals.
Time Frame: 14 days
Population: Parents and staff in SASEA Hub participating schools
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Control: School specific standard of COVID-19 care
Arm/Group | SASEA HUB | Control
Number analyzed (Participants) | 914 | 914
percentage of participants | 0.44 [0.41 to 0.48] | 0.40 [0.33 to 0.47]
Statistical Analysis 1: Comparison: SASEA HUB; Test type: Superiority; Mixed Models Analysis; Odds Ratio, log = 0.187, 95% CI 2-sided [-0.079 to 0.454], Standard Error of Mean 0.136

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the October to December only when schools were receiving the intervention. Adverse events were not monitored during the weeks where schools were receiving standard of care.
Description: 0 means - All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | SASEA HUB | Control
All-Cause Mortality (participants affected / at risk) | 0/917 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/917 | 0/0
Other Adverse Events (participants affected / at risk) | 0/917 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT05642000/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05642000/ICF_000.pdf